CLINICAL TRIAL: NCT02957318
Title: Effect of Potato Fiber on Appetite and Fecal Fat Excretion
Acronym: POFIBA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Anne Birgitte Raben, Professor, University of Copenhagen
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: B 326
Record Dates: First submitted 2016-11-01; First posted 2016-11-07 (Estimated); Last update posted 2017-09-13 (Actual); Status verified 2017-05

CONDITIONS: Fecal Fat Increased; Obesity; Appetite
MeSH Terms: conditions — Steatorrhea; Obesity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- FiberBind (Experimental)
  Interventions: Dietary Supplement: FiberBind
- RG-I fiber (Experimental)
  Interventions: Dietary Supplement: RG-I fiber
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: FiberBind — Potato pulp consisting of 68% fiber (5.5 soluble, 76.7% insoluble and 17.8% resistant starch), 9.7% water, 0.3% fat, 7.2% protein and 14% carbohydrates (starch).
  Arms: FiberBind
Dietary Supplement: RG-I fiber — Soluble fiber extracted from potato pulp consisting of 95% fiber and 5% water.
  Arms: RG-I fiber
Dietary Supplement: Placebo — Low-fiber control
  Arms: Placebo

SUMMARY:
Results have indicated that some dietary fibers increase fecal fat excretion and particularly viscous fibers suppress appetite sensation and reduce energy intake. Both these effects may contribute to body weight management.

Aim: The aim of the study is to investigate the potential of 3-weeks daily intake of potato pulp (FiberBind), rhamnogalacturonan I isolated potato fiber (RG-I) vs. a low-fiber control (placebo) on satiety and fecal fat excretion in healthy adults. Furthermore, a number of secondary endpoints are investigated.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Men
* BMI between 18.5 and 27.0 kg/m2
* Age 20-40 years

Exclusion Criteria:

* Intake of potatoes with main meals more frequent than 4 times per week
* Chronic diseases (known diabetes, cardiovascular disease, irritable bowels disease, colitis ulcerosa, crohn disease, or other chronic diseases which could affect the results of the present study)
* Gluten allergy
* Use of daily prescription medicine (mild analgesics are allowed)
* Use of lipid-lowering agents (e.g. Becel, HUSK)
* Use of food supplements of relevance to the study (such as pre- and probiotics)
* Irregular intake of vitamin /mineral supplements (two weeks prior to and during the entire study period)
* Smoking
* Elite athletes (>10 hours of strenuous physical activity per week)
* Blood donation (<1 month before study commencement and during study period)
* Participation in other clinical studies (<1 month before study commencement and during study period)
* Inability (physically or psychologically) to comply with the procedures required by the protocol judged by the Investigator

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2017-03-31 (Actual); Study Completion 2017-03-31 (Actual)

PRIMARY OUTCOMES:
Fecal fat excretion | Based on total feces collection the last 3 days of the 21-day intervention periods
Subjective appetite sensations | Assessed on 3-hour meal test on last day of the 21-day intervention periods
  Assessed by visual analogue scales (VAS)

SECONDARY OUTCOMES:
Ad libitum energy intake | Assessed 3 hours after intake of the test meal on last day of the 21-day intervention periods
Fecal energy excretion | Measured based on total feces collection the last 3 days of the 21-day intervention periods
Blood lipids (total cholesterol, HDL-cholesterol, LDL-cholesterol, triglycerides) | Measured before and after the 21-day intervention periods
Insulin and glucose | Measured before and after the 21-day intervention periods, and every 30 minutes during the 3-hour meal test on last day of the 21-week intervention periods
Gut permeability marker | Measured before and after the 21-day intervention periods
Gastric emptying rate (w. paracetamol) | Measured every 30 minutes during the 3-hour meal test on last day of the 21-day intervention periods
Gastrointestinal symptoms (questionnaire) | on day 1, 7, 14 and 22 of the 21-day intervention periods
Body weight | up to 21-day intervention periods
Blood pressure | up to 21-day intervention periods
Breath hydrogen | up to 21-day intervention periods
Gut microbiota | Measured in a fresh feces sample from day 19-21 of the intervention periods

CONTACTS AND LOCATIONS:
Locations (1):
- University of Copenhagen, Department of Nutrition, Exercise and Sports, Copenhagen, Denmark